CLINICAL TRIAL: NCT06045455
Title: The Importance of Multimodal CT Examination in Stroke Mimics Diagnosis: a Prospective Observational Multicenter Study
Brief Title: Multimodal CT Examination in Stroke Mimics Diagnosis
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); České Budějovice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NU23-04-00336; NU23-04-00336 (Other Grant/Funding Number: Ministry of Health of the Czech Republic); LM2023049 (Other Grant/Funding Number: STROCZECH, CZECRIN Large Research Infrastructure)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Stroke Mimics
Keywords: stroke mimics; neurological disorders; cerebrovascular accident; brain disorders; computer tomography; CT angiography; non-contrast head computed tomography; intravenous thrombolysis; National Institutes of Health Stroke Scale
MeSH Terms: conditions — Nervous System Diseases; Stroke; Brain Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neurological deficits (stroke or SM): All patients with acute neurological deficits (stroke or SM) will undergo neuroimaging diagnostic procedures initial multimodal brain CT (NCCT, CTP, CTA); then the follow-up NCCT within 24-36 hours.
  All patients without a confirmed concordant hypoperfusion or cerebral ischemia on their previous CT scans will undergo a magnetic resonance imaging (MRI) examination between the 3rd and 7th day after the admission to the hospital in order to confirm the diagnosis of SM.
  Interventions: Diagnostic Test: Multimodal brain CT; Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Multimodal brain CT — Multimodal brain CT includes NCCT, CTP, and CTA
Diagnostic Test: Magnetic resonance imaging (MRI) — MRI examination will be performed between the 3rd and 7th day after the admission to the hospital

SUMMARY:
The proposed project is a multicentre prospective observational clinical research focused on refining multimodal computer tomography (CT) diagnostics in stroke mimics. The main aim is to accurately identify SM in order to minimize the risk of receiving inappropriate treatment and possible development of complications, which can have a negative impact on the patient´s health. The project includes an analysis of pharmacoeconomic parameters. It will examine saved costs in the case of non-administration of unindicated treatment and it will compare the number of adverse events related to the administration of unindicated treatment in patients diagnosed with SM.

DETAILED DESCRIPTION:
The project has been designed as a prospective multicentre observational clinical research with applied outcomes leading to an improved provision of healthcare and healthcare costs. All patients older than 18 years admitted with suspected stroke will be included in the project.

The project will be implemented in 2 hospitals in the Czech Republic, namely the University Hospital in Ostrava and the Hospital in České Budějovice. The analyses will be performed at the University of Ostrava.

The primary objective of the project is to refine hospital diagnostics through the use of multimodal brain imaging (non-contrast CT (NCCT), CT angiography (CTA), and CT perfusion (CTP)) at hospital admission. The expected difference is at least 10% more patients with SM in the group diagnosed by the multimodal CT examination when compared to the group diagnosed with NCCT or NCCT/CTA. The primary objective is to demonstrate the specificity and sensitivity of multimodal brain imaging (NCCT, CTA, and CTP) when compared to the use of NCCT or NCCT/CTA in the acute diagnostics of SM in patients with a sudden focal neurological deficit (minimum 1 point on the National Institutes of Health Stroke Scale - NIHSS) within 24 hours from the onset of symptoms.

In addition to the importance of CTP in the diagnosis of stroke mimics, we will also analyze the significance of other clinical data.

The secondary objective is to compare the economic indicators and costs that will be saved by not providing inadequate treatment to patients with SM.

ELIGIBILITY:
Inclusion Criteria:

- an acute focal neurological deficit (minimum 1 point on the National Institutes of Health Stroke Scale - NIHSS) within 24 hours from the onset of symptoms

Exclusion Criteria:

* the last period of normality is unknown prior to multimodal CT examination
* the last period of normality is >24 hours prior to multimodal CT examination
* the diagnostic evaluation is incomplete
* a final neurologic diagnosis cannot be determined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients >18 years of age with an acute focal neurological deficit (minimum 1 point on the National Institutes of Health Stroke Scale - NIHSS) within 24 hours from the onset of symptoms will be enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The difference of patients with SM | up to 7 days
  The primary objective is to demonstrate the specificity and sensitivity of multimodal brain imaging (NCCT, CTA and CTP) when compared to the use of NCCT or NCCT/CTA in the acute diagnostics of SM in patients with a sudden focal neurological deficit (minimum 1 point on the National Institutes of Health Stroke Scale - NIHSS) within 24 hours from the onset of symptoms. The difference will be measured in per cent (%)

SECONDARY OUTCOMES:
Pharmacoeconomic analysis | 3 years
  The pharmacoeconomic analysis will include a Health Technology Assessment (HTA) in order to calculate the potential value of an innovation at an early stage, analysing not only the quality of life of patients, but also the costs associated with the treatment of stroke and SM. The calculation of costs is based on the average cost of thrombolysis and its associated treatment, representing the incremental cost (IC). Economic evaluation is organised as a test of dominance of improved results (meaning less complications associated with the administration of thrombolysis) and lower costs.
  In order to calculate the overall benefit, the value of the Quality of Life and the specific parameter of the Quality Adjusted Life Year (QALY) set for the Czech Republic will be used. The results will be reported as expected incremental costs (IC) and effects (E) expressed in quality-adjusted years of life (QALY).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Bar, prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (3):
- Czechia (3):
  - Hospital České Budějovice, České Budějovice, Jihočeský kraj
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Merino JG, Luby M, Benson RT, Davis LA, Hsia AW, Latour LL, Lynch JK, Warach S. Predictors of acute stroke mimics in 8187 patients referred to a stroke service. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):e397-403. doi: 10.1016/j.jstrokecerebrovasdis.2013.04.018. Epub 2013 May 13. PMID 23680681
- [Background] H Buck B, Akhtar N, Alrohimi A, Khan K, Shuaib A. Stroke mimics: incidence, aetiology, clinical features and treatment. Ann Med. 2021 Dec;53(1):420-436. doi: 10.1080/07853890.2021.1890205. PMID 33678099
- [Background] Vilela P. Acute stroke differential diagnosis: Stroke mimics. Eur J Radiol. 2017 Nov;96:133-144. doi: 10.1016/j.ejrad.2017.05.008. Epub 2017 May 5. PMID 28551302
- [Background] Siegler JE, Rosenberg J, Cristancho D, Olsen A, Pulst-Korenberg J, Raab L, Cucchiara B, Messe SR. Computed tomography perfusion in stroke mimics. Int J Stroke. 2020 Apr;15(3):299-307. doi: 10.1177/1747493019869702. Epub 2019 Aug 14. PMID 31409213
- [Background] Smajlovic D, Sinanovic O. Sensitivity of the neuroimaging techniques in ischemic stroke. Med Arh. 2004;58(5):282-4. PMID 15628251
- [Background] Austein F, Huhndorf M, Meyne J, Laufs H, Jansen O, Lindner T. Advanced CT for diagnosis of seizure-related stroke mimics. Eur Radiol. 2018 May;28(5):1791-1800. doi: 10.1007/s00330-017-5174-4. Epub 2017 Dec 7. PMID 29218615
- [Background] Shelly S, Maggio N, Boxer M, Blatt I, Tanne D, Orion D. Computed Tomography Perfusion Maps Reveal Blood Flow Dynamics in Postictal Patients: A Novel Diagnostic Tool. Isr Med Assoc J. 2017 Sep;19(9):553-556. PMID 28971638
- [Background] Ridolfi M, Granato A, Polverino P, Furlanis G, Ukmar M, Zorzenon I, Manganotti P. Migrainous aura as stroke-mimic: The role of perfusion-computed tomography. Clin Neurol Neurosurg. 2018 Mar;166:131-135. doi: 10.1016/j.clineuro.2018.01.032. Epub 2018 Jan 31. PMID 29414151
- [Background] Campbell BC, Weir L, Desmond PM, Tu HT, Hand PJ, Yan B, Donnan GA, Parsons MW, Davis SM. CT perfusion improves diagnostic accuracy and confidence in acute ischaemic stroke. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):613-8. doi: 10.1136/jnnp-2012-303752. Epub 2013 Jan 25. PMID 23355804
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Background] Van Cauwenberge MGA, Dekeyzer S, Nikoubashman O, Dafotakis M, Wiesmann M. Can perfusion CT unmask postictal stroke mimics? A case-control study of 133 patients. Neurology. 2018 Nov 13;91(20):e1918-e1927. doi: 10.1212/WNL.0000000000006501. Epub 2018 Oct 17. PMID 30333164
- [Background] Pohl M, Hesszenberger D, Kapus K, Meszaros J, Feher A, Varadi I, Pusch G, Fejes E, Tibold A, Feher G. Ischemic stroke mimics: A comprehensive review. J Clin Neurosci. 2021 Nov;93:174-182. doi: 10.1016/j.jocn.2021.09.025. Epub 2021 Sep 20. PMID 34656244
- [Derived] Dvornikova K, Kunesova V, Ely M, Ostry S, Cabal M, Reiser M, Machova L, Pavlinova M, Konde A, Elias P, Jonszta T, Havelka J, Volny O, Bar M. The importance of multimodal CT examination in stroke mimics diagnosis: design of prospective observational multicentre study. Front Neurol. 2024 Jun 4;15:1365986. doi: 10.3389/fneur.2024.1365986. eCollection 2024. PMID 38895699